CLINICAL TRIAL: NCT02942446
Title: Investigative Headgear With Nasal Pillows CPAP Mask
Brief Title: Investigative Headgear With Nasal Pillows Continuous Positive Airway Pressure (CPAP) Mask
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CIA 150
Record Dates: First submitted 2016-10-11; First posted 2016-10-24 (Estimated); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Headgear (Experimental): Investigative Headgear with CPAP mask
  Interventions: Device: Investigative Headgear with CPAP mask

INTERVENTIONS:
Device: Investigative Headgear with CPAP mask — Investigative Headgear with CPAP mask

SUMMARY:
This investigation is designed to evaluate the at-home usability, performance, user acceptance and reliability of the headgear with a CPAP mask for a duration of 6 months.

DETAILED DESCRIPTION:
20 participants will be recruited for the trial, consisting of male and female participants diagnosed with OSA and receiving CPAP or Bi-level Positive airway pressure (PAP) for the treatment of their Obstructive Sleep Apnea (OSA). These include current CPAP mask users.

ELIGIBILITY:
Inclusion Criteria:

* AHI≥5 from the diagnostic night
* ≥18 years of age
* Prescribed CPAP or Bi-level therapy for OSA
* Existing F&P Pilairo Q, Eson, Simplus mask users

Exclusion Criteria:

* Inability to give informed consent
* Patient intolerant to CPAP
* Anatomical or physiological conditions making CPAP therapy inappropriate
* History of respiratory disease or carbon dioxide (CO2) retention
* Pregnant or think they may be pregnant
* Investigated by Land Transport Safety Authority

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Reliability of the headgear using a Questionnaire | Monthly over a period of 6 months
  Assessment of headgear properties on a monthly basis via custom questionnaire via phone call
Durability of the headgear by testing | Monthly over a period of 6 months
  Assessment of headgear properties on a monthly basis, and changes to the headgear

SECONDARY OUTCOMES:
Performance in regards to leak of the headgear | Monthly over a period of 6 months
  Objective Leak Data (L/min) from the device download
Performance in regards to comfort of the headgear | Monthly over a period of 6 months
  Custom Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Gunson, BSc, Principal Investigator — Clinical Research Associate
Locations (1):
- Fisher & Paykel Healthcare, Auckland, New Zealand